CLINICAL TRIAL: NCT04882319
Title: An Evaluator-blinded, Randomized Within-subject Repeat Insult Study to Evaluate Potential Skin Irritation and Sensitization of HP-5000 (Diclofenac Sodium Topical System) in Healthy Adults
Brief Title: Irritation and Sensitization Study of HP-5000 Topical System
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Noven Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Noven Therapeutics (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-5000-US-06
Record Dates: First submitted 2021-05-03; First posted 2021-05-11 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Osteoarthritis of the Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HP-5000 Topical Patch (Experimental): HP-5000, placebo and saline will be administered simultaneously.
  Interventions: Drug: HP-5000 Topical Patch; Drug: HP-5000 Placebo Patch; Drug: Saline Patch

INTERVENTIONS:
Drug: HP-5000 Topical Patch — HP-5000, placebo and saline will be administered simultaneously
  Other Names: HP-5000 Patch
Drug: HP-5000 Placebo Patch — HP-5000, placebo and saline will be administered simultaneously
  Other Names: Placebo Control
Drug: Saline Patch — HP-5000, placebo and saline will be administered simultaneously
  Other Names: Saline Control

SUMMARY:
This study will assess skin irritation and sensitization for HP-5000 patch in healthy subjects.

DETAILED DESCRIPTION:
This is an evaluator-blinded, randomized phase 1 study evaluating skin irritation and sensitization of HP-5000 topical system in comparison to control patches. The study will consist of a 4-week Screening Phase and a Treatment Phase. The Treatment Phase will consist of the following periods: an Induction Period, a Rest Period followed by a Challenge Period and if needed, a Re-Challenge Period.

ELIGIBILITY:
Inclusion Criteria:

* Subject provides written informed consent prior to entering the study or undergoing any study procedures;
* Subject is a generally healthy male or female 18 to 65 years of age;
* Subject is considered to be healthy on the basis of medical history, physical examination, vital signs, normal electrocardiogram (ECG) and clinical laboratory test results.

Exclusion Criteria:

* Subject is pregnant or lactating, or females planning a pregnancy during the course of the trial;
* Subject has severe cardiac, renal or hepatic impairment;
* Subject has used any topical drugs at the patch application site within 72 hours prior to dosing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-06-03 (Actual); Primary Completion 2022-03-08 (Actual); Study Completion 2022-03-11 (Actual)

PRIMARY OUTCOMES:
Evaluating skin irritation with Mean Irritation Score (MIS) | 21 days
  To evaluate skin irritation after exposure to HP-5000, placebo and saline.
Evaluating skin sensitization with the number and proportion of subjects sensitized using descriptive statistics | 21 days
  To evaluate skin sensitization after exposure to HP-5000, placebo and saline.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Noven Pharmaceuticals, Inc.
Locations (1):
- TKL Research, Fair Lawn, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No